CLINICAL TRIAL: NCT00578396
Title: Phase I Biomarker Study of Dietary Grape-derived Low Dose Resveratrol for Colon Cancer Prevention
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Non applicable clinical trial
Sponsor: University of California, Irvine (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OCRT07046
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Colon Cancer
Keywords: Grapes and colon cancer prevention
MeSH Terms: conditions — Colonic Neoplasms | interventions — grp protein, Drosophila; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 (Active Comparator): 1 lb/day fresh red grapes
  Interventions: Dietary Supplement: grapes
- Dose Level 2 (Active Comparator): 2/3 lb/day fresh red grapes
  Interventions: Dietary Supplement: grapes
- Dose Level 3 (Active Comparator): 1/3 lb/day fresh red grapes
  Interventions: Dietary Supplement: grapes

INTERVENTIONS:
Dietary Supplement: grapes — 1 pound of seedless red grapes
  Other Names: dietary
  Arms: Dose Level 1
Dietary Supplement: grapes — 2/3 lb/day fresh red grapes
  Other Names: dietary
  Arms: Dose Level 2
Dietary Supplement: grapes — 1/3 lb/day fresh red grapes
  Other Names: dietary
  Arms: Dose Level 3

SUMMARY:
This study is designed to investigate the dietary influence of grapes in colon cancer prevention. A natural compound found in the skin of grapes, resveratrol, may protect against cancer by acting as an antioxidant (a chemical compound or substance that helps reduce damages due to oxygen). This compound is known to block colon cancer cell lines from growing in the laboratory. The purpose of this study is to determine the minimum amount of resveratrol-rich fresh red grapes needed to exhibit such signs of prevention.

DETAILED DESCRIPTION:
It has long been recognized that dietary factors influence the risk of developing colon cancer, with populations consuming a higher proportion of fruits and vegetables having lower risk. A compound found in the skin of grapes, resveratrol, has been purported to have colon cancer prevention activity though the dosages obtained through the diet have always seemed too low to produce inhibitory effects against cancer cells in the laboratory. We have found that low concentrations of resveratrol inhibit the Wnt pathway, a key signaling pathway which is activated in over 85% of colon cancers. We have also found in a small pilot trial that low dosages of freeze-dried grape powder can directly inhibit Wnt signaling in the normal colon and that grape powder was more effective than resveratrol alone in blocking Wnt throughput. This suggests that components of grapes may have direct activity in inhibiting a key signaling pathway and that this may correlate with cancer prevention activity.

In this study, we will directly test the impact of a diet containing a specific amount of red grapes in the context of a controlled amount of other resveratrol containing foodstuffs on Wnt signaling in the colon. This grape-supplemented diet provides a low-dose of resveratrol in conjunction with other potentially active components contained within the grapes. Participants will be normal volunteers and molecular studies will be done on colon tissue obtained by a limited flexible sigmoidoscopy before, and after, the red grape-containing diet is ingested. Different dosages of grapes will be utilized. This study will define the effect of dietary grape-derived low dose resveratrol on biomarkers related to the Wnt pathway, and provide critical information as to the utility of this nutritional approach toward colon cancer prevention.

For this study, seedless red grapes will be used. Ten participants will be enrolled at each dose level of grapes as follows:

* Dose level 1: 1 lb/day fresh red grapes
* Dose level 2: 2/3 lb/day fresh red grapes
* Dose level 3: 1/3 lb/day fresh red grapes

Participants will be normal volunteers identified through advertisements, referrals, and community outreach.

Primary Objective:

Define the minimum dietarily achievable amount of resveratrol-rich fresh red grapes which are effective in inhibiting Wnt signaling in human colonic mucosa.

Secondary Objectives

1. Define whether grape-supplemented diet affects colonic mucosa cell proliferation.
2. Define any side-effects associated with the resveratrol-rich dietary program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, male or female
* Participants must sign informed consent for enrollment
* Participants must have values for tests included in CBC, CMPAN and UA within normal range or no greater than 1.5x ULN or less than 0.75x LLN at prestudy to proceed to registration
* Participants must have normal limited flexible sigmoidoscopic examination on Day 15 to proceed to re-registration
* To receive Day 28 limited flexible sigmoidoscopy, participants must have taken >80% of prescribed dose of red grapes (based on food diary review)

Exclusion Criteria:

* Pregnant or lactating (and/or elevated ßHCG at enrollment)
* Known history of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Expression and cellular localization of beta-catenin in intestinal mucosa: localization of β-catenin. Expression of Wnt pathway target genes in intestinal mucosa: Wnt target gene expression | 2 yrs

SECONDARY OUTCOMES:
Define whether grape supplemented diet affects colonic mucosa cell proliferation. Ki67 staining method will be utilized on the pre- and post-resveratrol biopsy specimens. | 2 yrs
Define any side-effects associated with the resveratrol-rich dietary program. Laboratory testing is performed at specified timepoints in this protocol, along with history & physical, for the purposes of toxicity monitoring. | 2 yrs
Monitor resveratrol content of grapes throughout the course of the study. Grapes will be obtained from the same source as participants monthly throughout the study and the content of resveratrol will be measured. | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Randall F Holcombe, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States